CLINICAL TRIAL: NCT05265416
Title: Comparison Between the Effect of Piezocision and Low-level Laser Therapy on Patient-centered Outcomes in Patients Undergoing Upper Canine Retraction
Brief Title: Pain and Discomfort in Two Acceleration Methods of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-04-2022
Record Dates: First submitted 2022-02-14; First posted 2022-03-03 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Class II Malocclusion
Keywords: Piezosurgery; Diode laser; low-level laser; Pain
MeSH Terms: conditions — Overbite; Pain | interventions — Piezosurgery; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piezosurgery (Experimental): Piezocision will be applied in this group of patients using a piezosurgery knife.
  Interventions: Procedure: Piezosurgery
- Low-level laser therapy (Experimental): Low-level laser therapy will be applied in this group of patients using a diode laser device.
  Interventions: Other: Low-level laser therapy
- Traditional treatment (Active Comparator): No acceleration method will be performed in this group.
  Interventions: Device: Traditional treatment

INTERVENTIONS:
Procedure: Piezosurgery — Three vertical incisions will be made (3-mm depth and 8-10 mm length) after anesthesia. The cuts will be performed mesial and distal the upper canine as well as at an equal distance from the upper canine and 2nd premolar.
  Arms: Piezosurgery
Other: Low-level laser therapy — GaALAs diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) will be applied around the upper canine in 10 sites from buccal and palatal.
  Arms: Low-level laser therapy
Device: Traditional treatment — The canine retraction in this group will be performed in conventional method. Closed nickel-titanium coil springs applying 150 g of force per side will be used for retraction of the upper canine.
  Arms: Traditional treatment

SUMMARY:
54 patients who need extraction-based treatment of the maxillary first premolars with subsequent retraction of the maxillary canines will be divided randomly into three groups in this trial. The prolonged duration of the treatment period can cause many side effects such as white spots, caries, periodontal diseases, and pain and discomfort. So many efforts have been made to reduce the treatment time. Many procedures have been introduced to accelerate orthodontic tooth movement, which can category as surgical or non-surgical. Piezocision is a minimally invasive surgical method for accelerating orthodontic tooth movement and shortening treatment time. Low-level laser therapy (LLLT) is one of the physical acceleration methods that have contributed to decreasing treatment time.

There are three groups:

The first group (control group): the canine retraction in this group will be performed in conventional method.

The second group (Experimental group): the canine retraction in this group will be performed in association with piezocision.

The third group (Experimental group): the canine retraction in this group will be performed in association with low-level laser therapy.

DETAILED DESCRIPTION:
Closed nickel-titanium coil springs applying 150 g of force per side will be used for retraction of the upper canine.

Regarding the Piezocision, three vertical incisions will be made (3-mm depth and 8-10 mm length) after anesthesia. The cuts will be performed mesial and distal the upper canine as well as at an equal distance from the upper canine and 2nd premolar.

Regarding the low-level laser therapy (LLLT): GaALAs diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) will be applied around the upper canine in 10 sites from buccal and palatal. The middle of the extraction site will be also irradiated in 4 sites (2 buccally and 2 palatally). The LLLT will be applied 5 times in the first month of canine retraction. After that, until the class I canine relationship will be achieved, the irradiation will be repeated every two weeks.

The levels of pain and discomfort will be self-reported using a questionnaire with visual analog scales administered at five evaluation times during the first month of canine retraction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 17-28 years.
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. Patient had previous orthodontic treatment

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain | T1: after 24 hours of canine retraction commencement, T2: 3 days, T3: 7 days, T4: 14 days, and T5: 28 days following the commencement of the retraction.
  Assessment will be performed using questionnaires via Visual Analog scale.
Change in the levels of discomfort | T1: after 24 hours of canine retraction commencement, T2: 3 days, T3: 7 days, T4: 14 days, and T5: 28 days following the commencement of the retraction.
  Assessment will be performed using questionnaires via Visual Analog scale.
Change in the levels of swelling | T1: after 24 hours of canine retraction commencement, T2: 3 days, T3: 7 days, T4: 14 days, and T5: 28 days following the commencement of the retraction.
  Assessment will be performed using questionnaires via Visual Analog scale.
Levels of Eating difficulty | T1: after 24 hours of canine retraction commencement, T2: 3 days, T3: 7 days, T4: 14 days, and T5: 28 days following the commencement of the retraction.
  Assessment will be performed using questionnaires via Visual Analog scale.
Change in the levels of satisfaction | T5: 28 days following the commencement of the retraction.
  Assessment will be performed using questionnaires via Visual Analog scale and Two-point scale: (1) Yes (2) No.

CONTACTS AND LOCATIONS:
Overall Officials: Doa'a Tahseen Alfailany, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B, Latifeh Y. Evaluation of patient-centered outcomes associated with the acceleration of canine retraction by using minimally invasive surgical procedures: A randomized clinical controlled trial. Dent Med Probl. 2020 Jul-Sep;57(3):285-293. doi: 10.17219/dmp/120181. PMID 32909702
- [Background] Lombardo L, Ortan YO, Gorgun O, Panza C, Scuzzo G, Siciliani G. Changes in the oral environment after placement of lingual and labial orthodontic appliances. Prog Orthod. 2013 Sep 11;14:28. doi: 10.1186/2196-1042-14-28. PMID 24326120
- [Background] Aksakalli S, Calik B, Kara B, Ezirganli S. Accelerated tooth movement with piezocision and its periodontal-transversal effects in patients with Class II malocclusion. Angle Orthod. 2016 Jan;86(1):59-65. doi: 10.2319/012215-49.1. Epub 2015 May 19. PMID 25989211
- [Background] Keser E, Naini FB. Accelerated orthodontic tooth movement: surgical techniques and the regional acceleratory phenomenon. Maxillofac Plast Reconstr Surg. 2022 Jan 5;44(1):1. doi: 10.1186/s40902-021-00331-5. PMID 34984554
- [Background] Farid KA, Eid AA, Kaddah MA, Elsharaby FA. The effect of combined corticotomy and low level laser therapy on the rate of orthodontic tooth movement: split mouth randomized clinical trial. Laser Ther. 2019 Dec 31;28(4):275-283. doi: 10.5978/islsm.19-OR-19. PMID 32255919
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984